CLINICAL TRIAL: NCT02569840
Title: An Evaluation of the Tolerance and Acceptability of Neocate Junior an Amino Acid Based Formula for Children
Brief Title: Amino Acid Feed Children's Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NJ002
Record Dates: First submitted 2015-06-10; First posted 2015-10-07 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Milk Hypersensitivity
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amino Acid Feed (Other): An amino acid based multi-nutrient powdered feed
  Interventions: Dietary Supplement: Amino Acid Feed

INTERVENTIONS:
Dietary Supplement: Amino Acid Feed — Each child will receive the amino acid based feed for a period of up to 4 weeks (28 days). The feed prescription will be determined on an individual basis by the Dietitian responsible for the child's nutritional management. The child will take the feed orally or via a pre-existing naso-gastric, gastrostomy or jejunostomy tube.

SUMMARY:
This study of the tolerance and acceptability of an amino acid based feed will assess gastrointestinal (GI) tolerance, product intake and acceptability in relation to taste, smell, texture in 20 patients between 1-10 years currently using or requiring an amino acid based feed for the dietary management of Cows' Milk Allergy and food-allergy-associated conditions, over 4 weeks.

DETAILED DESCRIPTION:
Dietary management of Cows' Milk Allergy (CMA) involves avoiding cow's milk protein in the diet, whilst ensuring that an adequate nutritional intake is achieved with suitable alternative foods or prescribable feeds. A number of studies and clinical insights indicate that CMA is persisting longer than infancy, into later childhood and becoming more complex. If a child has CMA, eliminating the offending allergens whilst maintaining an intake of food that meets their nutritional requirements for growth and development is challenging due to the significant nutritional contribution these foods make to a child's diet, particularly milk and dairy products. This supports the need for alternatives to cow's milk to be available for children >1year of age to help meet their nutritional needs. Aminoacid based feeds are already widely used in clinical practice to meet this need. A new nutritionally complete amino acid based powdered feed for the dietary management of CMA, or other conditions where an amino acid based is recommended, in children aged 1-10yrs old, has been developed.

This study is to support the use of this new amino acid based feed in clinical practice. The study will evaluate the tolerance and acceptability of the amino acid based powdered feed in 20 children aged 1-10yrs of age receiving or requiring an amino acid based feed for the dietary management of CMA and food allergy associated conditions, over 4 weeks. The primary outcome will be gastrointestinal tolerance, with secondary outcomes of compliance, acceptability, nutrient intake and anthropometry.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 1-10 years
* Currently using or requiring an amino acid based feed
* Expected to receive at least 30% of their energy intake from the study product
* Written informed consent from parents / carer

Exclusion Criteria:

* Parenteral nutrition contributing more than 70% of total energy intake
* Children with major hepatic or renal dysfunction
* Participation in other studies within 2 weeks prior to entry of this study
* Investigator concern around willingness/ability of parent/carer to comply with protocol requirements

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Gastro intestinal tolerance questionnaire | 4 weeks
  Gastro-intestinal tolerance will be recorded at baseline and on days 1, 2, 3 and 7 of week 1 of the study. During weeks 2 and 3 tolerance will be recorded once at the end of each week on days 14 and 21. During week 4, tolerance will be recorded on days 26, 27 and 28. Tolerance will be recorded using a standardised gastro-intestinal tolerance questionnaire, to be completed by the parents/carer

SECONDARY OUTCOMES:
Compliance with feed prescription (amount prescribed versus consumed) | 4 weeks
  Compliance with feed prescription will be assessed daily throughout the study by recording how much feed was received, to be recorded by the parents/carer. The amount prescribed by the Dietitian will be recorded at the start of the study, and any changes to this prescription also noted
Product acceptability questionnaire | 4 weeks
  Feed acceptability (ease of use) will be assessed at the end of week 4 by questionnaire completed by the parents/carer.
Nutrient intake (energy, protein and micronutrients) | 4 weeks
  Nutrient intake, including the intake of all nutrition provided (including the study product, any parenteral feeding, other enteral tube feeding, foods, drinks etc) will be recorded at baseline and on Day 28 by the Dietitian using 24hour recall, and then in 3 day food diaries at baseline (Days 1, 2 and 3) and Week 4 (Days 26, 27 and 28) by the parent/carer. A dietary analysis program will be used to calculate total dietary intake
Weight (kg) | 4 weeks
  For safety purposes, at baseline and at the end of week 4, body weight (kg) will be measured where possible using standard methods, to the nearest 0.1kg using a weighing scale without heavy clothing. Height will also be measured, wherever possible, using standard measures to the nearest 0.1cm. For children up to 2yrs of age, head circumference will be measured where possible, using standard methods to the nearest 0.1cm
Height (cm) | 4 weeks
  For safety purposes, at baseline and at the end of week 4, body weight (kg) will be measured where possible using standard methods, to the nearest 0.1kg using a weighing scale without heavy clothing. Height will also be measured, wherever possible, using standard measures to the nearest 0.1cm. For children up to 2yrs of age, head circumference will be measured where possible, using standard methods to the nearest 0.1cm
Head circumference (cm) | 4 weeks
  For safety purposes, at baseline and at the end of week 4, body weight (kg) will be measured where possible using standard methods, to the nearest 0.1kg using a weighing scale without heavy clothing. Height will also be measured, wherever possible, using standard measures to the nearest 0.1cm. For children up to 2yrs of age, head circumference will be measured where possible, using standard methods to the nearest 0.1cm
Safety by Adverse Event reporting | 4 weeks
  All adverse events will be recorded, throughout the study.

IPD SHARING:
Plan to Share IPD: No